CLINICAL TRIAL: NCT04677608
Title: An Italian Multicenter Prospective Study on Pulmonary Hypertension Modality of Death and Validation of Reveal Risk Score
Brief Title: Pulmonary Hypertension Modality of Death and Validation of REVEAL Risk Score
Acronym: ASPYRE-1
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: iPHNET (italian Pulmonary Hypertension NETwork) (Other)
Responsible Party: Sponsor
Other Study IDs: ASPYRE-1
Record Dates: First submitted 2020-12-16; First posted 2020-12-21 (Actual); Last update posted 2020-12-21 (Actual); Status verified 2020-12

CONDITIONS: Pulmonary Arterial Hypertension
MeSH Terms: conditions — Pulmonary Arterial Hypertension

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Pulmonary Arterial Hypertension (PAH) is a chronic disease characterized by a progressive increase in pulmonary vascular resistance (PVR), which leads to right ventricular (RV) failure, and ultimately death.

Different studies have outlined how various factors as vascular resistance, functional class, age, correlate with mortality. However, the modality of death and risk factors for mortality in patients with PAH are little known. For this purpose, more studies are necessary to analyze the risk factors related to modality of death in PAH.

DETAILED DESCRIPTION:
Pulmonary Arterial Hypertension (PAH) is a disease characterized by dyspnea, fatigue, chest pain, and syncope. PAH results from a narrowing of the small arteries and arterioles, resulting in elevation of pulmonary vascular resistance and leading to the development of right ventricular failure and death if untreated. Worldwide, it is estimated that between 130,000 and 260,000 persons have PAH. Mean age at diagnosis is 35 years, and most patients present with moderate-to-severe disease. PAH occurs most often in otherwise healthy persons, and more often in women than men. There is no known cure for PAH, and the goal of current therapy is to control symptoms of the disease and hopefully slow its progression. Prognosis is poor in patients with PAH, and is similar to that of many advanced cancers; five-year survival in the absence of treatment is only about 50%.

Comparatively little is known about the modality of death and risk factors for mortality in patients with PAH. In a recent systematic review, a little consensus was found among the 54 studies identified, most of which involved relatively few patients.

Of 107 risk factors that were found to be significantly related to mortality in at least one study, only 10 demonstrated "a reproducible predictive association with mortality." Benza and colleagues recently reported on a retrospective analysis of information from 2716 PAH patients enrolled in the US Registry to Evaluate Early and Long-Term PAH Disease Management (REVEAL). This study was much larger than any previous one and too recent to be included in the aforementioned systematic review. In multivariate analysis, they found that high pulmonary vascular resistance (PVR >32 Wood Units), PAH secondary to portal hypertension, NYHA Functional Class IV, male gender, older age (>60 years), and family history of PAH were all predictive of 1-year mortality. Interestingly, none of the 107 risk factors identified in the systematic review concerned nutritional status (e.g., body mass index [BMI], serum albumin). Preliminary results from an ongoing European study, however, suggest that low BMI is an important independent predictor of mortality in patients with PAH, possibly including death due to chronic heart failure, sudden cardiac death, and/or death due to extracardiac causes. If this is indeed the case, then improvements inpatient nutrition may offer the potential to extend life expectancy at the relatively low burden and minimal cost.

Given current uncertainty about the mode of death and risk factors for mortality in PAH, a new study is planned to examine this issue, with a particular focus on the independent contribution of BMI as a risk factor for mortality.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of PAH (group 1) according to ESC/ERS classification

Exclusion Criteria:

* Diagnosis of one of the following groups of PH:
* Group 1: PAH associated with congenital heart disease
* Group 2: PH due to left heart disease
* Group 3: PH due to lung disease and/or hypoxia
* Group 4: Chronic Thromboembolic PH (CTEPH)
* Group 5: PH due to miscellaneous causes

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects with a confirmed diagnosis of Pulmonary Hypertension (PH) by Right Heart Catheterization (RHC), according to pre-capillary pulmonary hypertension (mPAP ≥ 25mmHg, PCWP ≤15 mmHg, PVR > 3 WU)
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2020-07-21 (Actual); Primary Completion 2021-04-30 (Estimated); Study Completion 2022-08-31 (Estimated)

PRIMARY OUTCOMES:
Modality of death | two years
  to identify the different modality of death in patients with PAH
Risk factors | two years
  to identify risk factors for mortality in patients with PAH

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Clinical, Internal, Anesthesiological and Cardiovascular Sciences. AOU Policlinico Umberto I, Rome, Italy